CLINICAL TRIAL: NCT06751810
Title: EVALUATION OF A NEW SUPPLEMENT ON NUTRITIONAL STATUS IN CHILDREN WITH FOOD ALLERGY
Brief Title: Nutritional Status in Children With Food Allergy: Evaluation of a New Supplement
Acronym: ALLERGYSTOP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Md, PhD, Principal Investigator, Federico II University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 09/24
Record Dates: First submitted 2024-12-15; First posted 2024-12-30 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2024-12

CONDITIONS: Food Allergies
Keywords: allergy; food allergy; cow milk protein allergy
MeSH Terms: conditions — Food Hypersensitivity; Hypersensitivity | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplement (Experimental): Subjects assigned to receive the treatment
  Interventions: Dietary Supplement: Food supplement
- Placebo (Placebo Comparator): Subjects assigned to receive the placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Food supplement — The nutritional composition of the food supplement comprises:
  sodium butyrate, inactivated Lactobacillus rhamnosus GG Perilla frutescens dry extract quercetin fructo-oligosaccharides Vitamin D3 omega 3 polyunsaturated acids
  Arms: Supplement
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Allergic diseases are rising globally. By 2025, over half of the European population is projected to be affected by some form of allergy, with the highest rates among infants and young children. This growing prevalence also has a significant economic impact, resulting in more than 100 million lost work and school days each year due to allergic conditions.

Allergies arise from a breakdown in immune tolerance mechanisms. Current research suggests that the development is influenced by genetic, environmental, and gene-environment interactions, leading to immune system dysfunction, partly mediated by epigenetic mechanisms. Various factors have been proposed as contributors to FA onset. Among the unchangeable risk factors are male sex, race/ethnicity (with higher risks among Asian and Black children compared to White children), and genetics (familial associations, HLA, and specific genes).

Modifiable risk factors also play a role, with growing evidence showing that environmental influences, such as the use of antibiotics, antiseptic agents, and a high-fat, low-fiber diet, negatively affect microbiome composition. Additional risk factors potentially affecting FA onset include atopic diseases (such as comorbid atopic dermatitis), increased hygiene, vitamin D deficiency, reduced consumption of omega-3 polyunsaturated fatty acids and antioxidants, the use of antacids (which hinder the digestion of allergens), obesity, and the timing and route of food exposure (increased risk with delayed oral ingestion of allergens coupled with environmental exposure). The microbiome also plays a critical role in these processes.

Currently, no Food and Drug Administration (FDA)-approved treatment exists for FA, and the standard approach is strict dietary avoidance of the triggering allergens. As a result, the nutritional burden of elimination diets can be substantial, leading to risks such as growth failure, micronutrient deficiencies, and feeding challenges with long-term consequences.

ELIGIBILITY:
Inclusion Criteria:

* subjects with food allergy
* Gestational age ≥ 37 weeks

  * Stable clinical condition and free from any symptoms possibly related to food allergy at least four weeks prior to study enrollment
  * Observing a strict cow's milk elimination diet for at least 4 weeks prior to study enrollment and until the completion of the study
  * Parent(s) or legal guardian agrees not to enroll infant or child in another interventional clinical study while participating in this study
  * Written informed consent obtained from at least one parent (or legally acceptable representative [LAR], if applicable)
  * Infant or child's parent(s) / LAR is of legal age of majority, must have parental authority, must understand the informed consent form and other study documents, and are willing and able to fulfill the requirements of the study protocol

Exclusion Criteria:

* other concomitant diseases
* Infant or child's parent has other medical or psychiatric condition that, in the judgement of the Investigator, would make the infant or child inappropriate for entry into the study.
* Currently participating or having participated in another interventional clinical study within 4 weeks prior to enrollment.

Ages: 36 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-12-30 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
body growth parameters | after 6 months of treatment
  body mass index

SECONDARY OUTCOMES:
biochemical values | after 6 months of treatment
  serum vitamin D levels
biochemical values | after 6 months of treatment
  serum DHA levels
Cytokines production | after 48 days
  Th2 cytokines (IL-4, IL-5, IL-13), IL-10 production
regulatory T cells (Tregs) production | after 4 days
  regulatory T cells (Tregs)
regulatory dendritic cell markers production | after 4 days
  regulatory dendritic cell markers (Tgfb1, Ifna2, Ptgs2, Csf2)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Traslational Medical Science - University of Naples Federico II, Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: No